CLINICAL TRIAL: NCT05007249
Title: Benefit of the Chalaxie Pedagogical Tool in the Management of Overweight or Obese Children With Intellectual Disability : a Pilot Monocentric Prospective Study.
Acronym: CHALAXIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GHR 1169
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2021-08

CONDITIONS: Pediatric Obesity
Keywords: intellectual disability; patient therapeutic education; pedagogical evaluation
MeSH Terms: conditions — Pediatric Obesity; Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overweight or obese minors with intellectual disability (Other)
  Interventions: Procedure: Use of the Chalaxie pedagogical evaluation tool

INTERVENTIONS:
Procedure: Use of the Chalaxie pedagogical evaluation tool — Use of the Chalaxie pedagogical evaluation tool during two visits

SUMMARY:
The main objective of this study is to determine the benefit of the Chalaxie pedagogical evaluation tool in the management of overweight or obese children with intellectual disability.

Chalaxie is a software developped as a pedagogical evaluation tool. It is used in the therapeutic education of overweight and obese children and allow the clinican to explore several skills of the child, such as self-esteem.

DETAILED DESCRIPTION:
Secondary objectives

1. To assess the feasibility of the Chalaxie tool use during a medical visit;
2. To assess the relevance of the Chalaxie tool for the pediatrician;
3. To describe the characteristics of the patients followed at the "Réseau ODE";
4. To evaluate patient self-esteem.

Conduct of research After receiving written consent from the study participant and parental authority, the patients will have two visits with the pediatrician during which they will use the Chalaxie pedagogical evaluation tool. At the first visit, they will use the self-esteem assessment module. At the second visit (i.e. final visit), which should take place between 3 weeks and 2 months after the first visit, they will use a module of their choice.

ELIGIBILITY:
Inclusion Criteria:

* Minor patient of 11 years of age or older
* Overweight or obese patient respectively defined as a BMI ≥ IOTF 25 and ≥ IOTF 30
* Mild intellectual disability defined as intelligence quotient (IQ) ≥ 55 and <70 or (if IQ unknown) patient in a special education institution (ULIS, IM-PRO)
* Affiliated or beneficiary of a social security scheme
* Written consent of the patient and one of the parental authority holder

Exclusion Criteria:

* Patient with a severe autistic disorder
* Patient who already used the Chalaxie tool during his/her follow-up
* Difficulties in understanding the instructions for using the software and/or difficulties in using a computer

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Self-report patient perception questionnaire | through study completion, an average of 2 months
  The benefit of the Chalaxie pedagogical evaluation tool will be measured with the patient perception questionnaire completed at the final visit. It consists of seven single choice questions and one open question.

SECONDARY OUTCOMES:
Duration of the visit | on enrollment day only
  Duration will be measured from the moment the written consent is obtained until the end of the visit
Duration of the use of the self-esteem assessment module | on enrollment day only
  Duration will be measured from the moment the investigator clicks on the module until the completion of the last question.
Clinician perception questionnaire | Through study completion, on enrollment day to the final visit, an average of 2 months
  Clinician perception questionnaire consists of 12 single choice questions.
Self-esteem | on enrollment day only
  Self-esteem will be evaluated with the self-esteem assessment module. It consists of 6 questions with a visual scale of 6 emoticons. It also includes a 4-modality question assessing overall self-esteem that is completed by the patient and pediatrician respectively.

CONTACTS AND LOCATIONS:
Overall Officials: fatiha Guemazi-Kheffi, MD, Principal Investigator — Groupe Hospitalier de la Région de Mulhouse et Sud-Alsace
Locations (1):
- Hôpital Emile Muller (GHRMSA), Mulhouse, France

IPD SHARING:
Plan to Share IPD: No